CLINICAL TRIAL: NCT00002130
Title: A Long-Term, Follow-On Safety Study of Four Doses of OPC-8212 (Vesnarinone) in HIV-Infected Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 234C; 22-93-253
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antiviral Agents; vesnarinone
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vesnarinone

INTERVENTIONS:
Drug: Vesnarinone

SUMMARY:
To examine the continued safety and tolerability of four doses of vesnarinone in HIV-infected patients who have completed a short-term study (less than 12 months on continuous treatment) of the drug.

DETAILED DESCRIPTION:
Patients who have completed a limited duration study (less than 12 months of continuous treatment) of vesnarinone on protocols FDA 234A or FDA 234B and who have no current signs or symptoms of AIDS-defining illnesses may roll over to this study and continue receiving their regimen of vesnarinone for 12 months beyond their original participation.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii, candida, and mycobacteria.
* Acyclovir for acute treatment of herpes.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antiretroviral agents, including ddI, ddC, AZT, and d4T.
* Immunosuppressive agents.
* Investigational HIV drugs/therapies including vaccines.
* Interferon or other immunomodulating agents.
* Corticosteroids (other than topical).
* Megestrol acetate.
* Agents known to cause neutropenia.
* Ganciclovir.
* Cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

* Poor compliance (less than 80 percent of drug taken) on the Phase I protocol (FDA 234A or FDA 234B).
* Missed more than one clinic visit on the Phase I protocol.

Prior Medication:

Excluded:

* Acyclovir as prophylaxis for herpes within 48 hours prior to study entry.

Patients meet the following criteria:

Successful completion of short-term therapy with vesnarinone on FDA 234A or FDA 234B.

Active illicit drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA School of Medicine, Los Angeles, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia